CLINICAL TRIAL: NCT06550284
Title: Small Nerve Fiber Activity in Patients with Carpal Tunnel Syndrome Assessed Via Quantitative Sensory Testing
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brooke Army Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Cortney Shewmaker, Orthopedic Manual Physical Therapy Fellow, Brooke Army Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C.2024.041
Record Dates: First submitted 2024-08-09; First posted 2024-08-13 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Carpal Tunnel Syndrome
Keywords: carpal tunnel syndrome; quantitative sensory testing; median nerve; neuropathy; small nerve fiber
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — Physical Therapy Modalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Carpal Tunnel Syndrome (Experimental): Age 18-65 years with unilateral carpal tunnel syndrome.
  Interventions: Other: Physical Therapy

INTERVENTIONS:
Other: Physical Therapy — The intervention will be physical therapy standard care.

SUMMARY:
The diagnosis of carpal tunnel syndrome (CTS) is typically based on clinical findings and confirmatory electrodiagnostic testing. However, electrodiagnostic testing can only assess large A-alpha and A-beta nerve fibers. Quantitative sensory testing (QST) is a series of tests used to assess small nerve fiber changes in the A-delta, c-fibers, and A-beta nerve fibers as well. Previous studies have used QST to assess small nerve fiber changes related to carpal tunnel syndrome and found changes compared to controls. This study will utilize a course of standard physical therapy care and assess for any changes to small nerve fiber activity and how those changes may or may not relate to patient outcomes.

DETAILED DESCRIPTION:
Purpose: To assess changes in A-beta, A-deta, and C-fiber function after standard physical therapy interventions in individuals with CTS.

Specific Aim 1 (primary aim): Determine if A-beta, A-deta, and C-fiber functions change following a course of Physical Therapy (PT) in individuals with CTS.

Specific Aim 2 (secondary aim): Describe the relationship between changes in QST and changes in a patient-reported outcome measure after a course of PT in individuals with a clinical diagnosis of CTS.

Specific Aim 3 (secondary aim): Determine if there are differences in A-beta, A-deta, and C-fiber function between the affected and unaffected wrists in individuals with a clinical diagnosis of CTS.

ELIGIBILITY:
Inclusion Criteria:

DEERS eligible Age 18-65 Pain and paresthesia in the median nerve distribution A positive Phalen test A positive Tinel test over the carpal tunnel Willing to attend physical therapy

Exclusion Criteria:

Nerve root signs consistent with a radiculopathy Suspected radial and ulnar nerve involvement based on monofilament testing Bilateral CTS Previous hand surgery Injections in the upper quarter in the last 6 months Cervical, shoulder, or UE trauma in the last 6 months Currently pregnant or postpartum within the last 6 months No more than minimal care (evaluation and patient education, 1 visit) for the current episode

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-11-12 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Quantitative Sensory Testing (QST) | From enrollment until the end of the study at 12 weeks
  QST is a test method that measures sensory thresholds for temperature sensations, touch, vibration, and pain and is described in section 10.1. All thermal testing (CDT, WDT, CPT, and HPT) will be performed via the TSA 2 Thermosensory Stimulator.

SECONDARY OUTCOMES:
Boston Carpal Tunnel Questionnaire (BCTQ) | From enrollment until the end of the study at 12 weeks
  The BCTQ is a self-based outcome scale measured with 2-parts, the symptom severity scale and functional status scale. Both scales are likert scales 1-5.
Numeric Pain Rating Scale (NPRS) | From enrollment until the end of the study at 12 weeks
  he NPRS is an 11-point scale ('0' indicating no pain, and '10' worst imaginable pain) that will be used to assess pain intensity. This will be measured as the mean of three pain ratings: best pain rating over 24 hours, worst pain rating over 24 hours, and current pain rating.

CONTACTS AND LOCATIONS:
Locations (1):
- Brooke Army Medical Center, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided
Requests for deidentified data will be considered on a case by case basis.